CLINICAL TRIAL: NCT05054296
Title: Modifying Metabolic Syndrome and Cardiovascular Risk for Prostate Cancer Patients on ADT Using a Supervised Exercise Program and Continuous Fitbit Monitoring
Brief Title: Modifying Metabolic Syndrome and Cardiovascular Risk for Prostate Cancer Patients on ADT Using a Risk Factor Modification Program and Continuous Fitbit Monitoring
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0938; NCI-2019-08624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0938 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-01-06; First posted 2021-09-23 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (education exercise packet, FitBit) (Active Comparator): Patients receive general education exercise packet with instruction to exercise regularly for up to 150 minutes weekly. Patients also wear a FitBit daily over 16 weeks.
  Interventions: Behavioral: Educational Intervention; Device: FitBit; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (exercise program FitBit) (Experimental): Patients participate in supervised and self-directed exercise sessions over 60 minutes BIW for up to 16 weeks. Patients also wear a FitBit daily over 16 weeks.
  Interventions: Behavioral: Exercise Intervention; Device: FitBit; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Educational Intervention — Receive general education exercise packet
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (education exercise packet, FitBit)
Behavioral: Exercise Intervention — Participate in supervised and self-directed exercise sessions
  Arms: Group II (exercise program FitBit)
Device: FitBit — Wear FitBit for activity tracking
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well an exercise program and continuous Fitbit monitoring work for managing metabolic syndrome and cardiovascular disease risk in patients with prostate cancer that has spread to other places in the body (metastatic) or has come back (recurrent) and does not response to treatment (refractory) and are receiving androgen deprivation therapy. Balancing treatment efficacy, drug side effects, and competing comorbidities with prostate cancer is essential. This trial is being done to learn if an exercise program can help to improve metabolic syndrome and cardiovascular (heart) fitness in prostate cancer patients who are receiving androgen deprivation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the relationship between a 16-week exercise program with continuous Fitbit monitoring and cardiovascular fitness (defined by change in 10-year atherosclerotic cardiovascular disease [ASCVD] risk score), as compared to Fitbit monitoring alone, in prostate cancer patients on androgen deprivation therapy (ADT).

SECONDARY OBJECTIVES:

I. Determine the length of cardiovascular fitness effect (measured using 10-year ASCVD risk 12 weeks post intervention) for a 16-week exercise program with continuous Fitbit monitoring in prostate cancer patients on ADT.

II. Screen for a relationship between a 16-week exercise program with continuous Fitbit monitoring and metabolic syndrome severity (defined by change in metabolic severity index z-score), as compared to Fitbit monitoring alone, in prostate cancer patients on ADT.

III. Measure the relationship between the exercise intervention and prostate-specific antigen (PSA) velocity, compared to Fitbit monitoring alone.

IV. Measure the relationship between the exercise intervention and physical fitness (using V02 and body composition), compared to Fitbit monitoring alone.

V. Measure the relationship between the exercise intervention and physical activity (step count)/heart rate, compared to Fitbit monitoring alone.

VI. Measure the relationship between the exercise intervention and physical activity (as measured by the Godin Leisure Time Physical Activity Questionnaire) compared to Fitbit monitoring alone.

VII. Measure the relationship between the exercise intervention and, quality of life/symptom burden, compared to Fitbit monitoring alone (measured by the following patient reported surveys: National Cancer Institute-patient reported outcomes-Common Terminology Criteria for Adverse Events [NCI-PRO-CTCAE], Patient Reported Outcomes Measurement Information System [PROMIS] Fatigue and Physical Function, Self Efficacy, European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire Core30 [QLQ-C30] and Prostate Cancer 25 [PR25]).

EXPLORATORY OBJECTIVE:

I. Explore the relationship between the exercise intervention and markers of insulin resistance, inflammation/immune function and metabolism utilizing pre- and post-intervention peripheral blood analysis.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive general education exercise packet with instruction to exercise regularly for up to 150 minutes weekly. Patients also wear a FitBit daily over 16 weeks.

GROUP II: Patients participate in supervised and self-directed exercise sessions over 60 minutes twice a week (BIW) for up to 16 weeks. Patients also wear a FitBit daily over 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Presence of metastatic disease documented on imaging studies (bone scan, computed tomography [CT] and/or magnetic resonance imaging [MRI]) or biochemical recurrence/refractoriness following local therapy (prostatectomy or radiation)
* Stable or improving disease activity as demonstrated by stable or improving PSA over at least 2 months
* On gonadotropin-releasing hormone (GnRH) agonist or GnRH antagonist or status post-surgical castration for at least 3 months
* Combination ADT with abiraterone or enzalutamide is permitted
* Anticipation to remain hypogonadal for at least 6 months subsequently
* Asymptomatic bone metastasis is permissible (exercise will be modified and patients monitored)
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients must be able to finish a maximal exercise stress test which will be assessed by cardiopulmonary exercise testing using a standardized protocol ^70 supervised by a cardiologist
* Hemoglobin >= 9.0 g/dL independent of transfusion and/or growth factors within 3 months prior to enrollment
* Platelet count >=75,000/uL independent of transfusion and/or growth factors within 3 months prior to enrollment
* Access to a smart phone with android or iPhone OS (iOS) operating systems
* Able to speak and comprehend English

Exclusion Criteria:

* Current use of any other systemic therapy for prostate cancer with the exception of gonadotrophin releasing hormone (GnRH) agonists/antagonists, abiraterone, enzalutamide, bisphosphonates or RANK-ligand inhibitors (for bone metastases) which are allowed
* Any underlying comorbid medical or psychiatric condition, which in the opinion of the Investigator, will make participation in our exercise intervention hazardous or obscure the interpretation of adverse events
* Inability to walk 400 meters or undertake upper and lower limb exercise, and resistance training in the previous 3 months
* Chemotherapy treatment within 28 days of study enrollment
* Symptomatic bone metastasis
* Any investigational pharmaceutical products
* Radiation therapy or surgical intervention for prior bone metastasis
* Clinically significant active malignancy other than prostate cancer
* Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (>= 450 m/sec)
* Clinically significant heart disease that may impact safety of independent or supervised exercise including preexisting coronary artery disease, myocardial infarction or arterial thrombotic events in the past 6 months, severe or unstable angina, history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsade de pointes), New York Heart Association Class III-IV heart disease or cardiac ejection fraction measurement of < 40% at baseline
* Untreated symptomatic spinal cord compressions
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Atherosclerotic cardiovascular disease (ASCVD) 10-year risk score | Through the study completion, an average of a year.
  The 16-week exercise program would affect this risk score through reduction of systolic blood pressure (SBP) and cholesterol while increasing high-density lipoprotein (HDL).
  · A 0 to 4.9 percent risk is considered low. Eating a healthy diet and exercising will help keep your risk low.
  Medication is not recommended unless your LDL, or "bad" cholesterol, is greater than or equal to 190.
  * A 5 to 7.4 percent risk is considered borderline. Use of a statin medication may be recommended if you have certain conditions, or "risk enhancers." These conditions may increase your risk of a heart disease or stroke. Talk with your primary care provider to see if you have any of the risk enhancers in the list below.
  * A 7.5 to 20 percent risk is considered intermediate. It is recommended that you start with moderate-intensity statin therapy.
  * A greater than 20 percent risk is considered high. It is recommended that you start with high-intensity statin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Logothetis, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org